CLINICAL TRIAL: NCT00939822
Title: Statin Effects on Beta-Amyloid and Cerebral Perfusion in Adults at Risk for AD: "Statins in Healthy, At-Risk Adults: Impact on Amyloid and Regional Perfusion (SHARP)" Study
Brief Title: Statin Effects on Beta-Amyloid and Cerebral Perfusion in Adults at Risk for Alzheimer's Disease
Acronym: SHARP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2015-0038; R01AG031790-01A1 (NIH); H-2009-0030 (Other: Old IRB Number); H-2008-0275 (Other: Old IRB Number)
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Results first posted 2019-08-09 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Simvastatin (Experimental): 40 mg. Simvastatin/day
  Interventions: Drug: Simvastatin
- Placebo (Placebo Comparator): Matching Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Simvastatin — 40 mg Simvastatin/day
  Arms: Simvastatin
Drug: Placebo — Matching Placebo
  Arms: Placebo

SUMMARY:
The purpose of the research is to see how simvastatin affects a substance in the body called beta-amyloid. Beta-amyloid is found in the brain and in the liquid around the brain and spinal cord. High amounts of beta-amyloid may be associated with a greater risk of getting Alzheimer's disease. This study will see if simvastatin can lower the amount of beta-amyloid in the spinal fluid. This study will also see if simvastatin affects memory and thinking, blood flow in the brain, and blood vessel function. The investigators hope that future studies show whether simvastatin might prevent memory loss and decrease the chance of developing Alzheimer's disease.

DETAILED DESCRIPTION:
Studies show that some medicines that lower cholesterol may reduce the risk of developing Alzheimer's disease, but this has not yet been proven in humans. We are looking for individuals to participate in this study to see if a cholesterol-lowering medication, called simvastatin affects blood flow to the brain, blood vessel function and a substance in the spinal fluid related to the changes in Alzheimer's disease.

The SHARP study included 88 adults ages 40-72 with parental history of documented Alzheimer's disease. The study had 9 visits over the course of 18 months. Participants had fasting blood tests collected, completed a medical history questionnaire and medication side effect review, underwent lumbar puncture procedure, completed memory testing, and had ultrasound and MRI procedures. Participants were randomly assigned to receive either simvastatin or a placebo each night for 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Parent diagnosed with Alzheimer's disease
* Age 40-72

Exclusion Criteria:

* Active liver disease
* History of adverse reaction to statins
* Contraindication to lumbar puncture
* Elevated creatine kinase and creatinine lab values
* Use of medications known to interact with statins
* History of dementia or mild cognitive impairment
* Currently pregnant or planning to become pregnant
* Use of large quantities of grapefruit juice (more than 1 quart per day)
* Contraindications to MRI (for MRI sub-study)
* Currently on cholesterol-lowering medication or use in past 4 months
* History of heart attack, heart problems, stroke and/or diabetes
* Drinking more than a quart of grapefruit juice per day
* Metal implants, or metal debris in body (MRI)
* List of medications that interact with simvastatin

Ages: 40 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2009-03 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia M. Carlsson, MD, MS, Principal Investigator — UW Madison School of Medicine and Public Health
Locations (1):
- Karen Lazar, Fitchburg, Wisconsin, United States

REFERENCES:
- [Derived] Vogt NM, Hunt JFV, Ma Y, Van Hulle CA, Adluru N, Chappell RJ, Lazar KK, Jacobson LE, Austin BP, Asthana S, Johnson SC, Bendlin BB, Carlsson CM. Effects of simvastatin on white matter integrity in healthy middle-aged adults. Ann Clin Transl Neurol. 2021 Aug;8(8):1656-1667. doi: 10.1002/acn3.51421. Epub 2021 Jul 18. PMID 34275209
- [Derived] Gepner AD, Lazar K, Hulle CV, Korcarz CE, Asthana S, Carlsson CM. Effects of Simvastatin on Augmentation Index Are Transient: Outcomes From a Randomized Controlled Trial. J Am Heart Assoc. 2019 Oct 15;8(20):e009792. doi: 10.1161/JAHA.118.009792. Epub 2019 Oct 12. PMID 31607205
- See also: Related Info — http://wisconsinadrc.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Asymptomatic middle-aged adults (ages 40-72 years) with parental history of AD were recruited from the community through local memory clinics, newsletters, educational talks, booths at health fairs, and newspaper and magazine advertisements.
Pre-assignment Details: Screened individuals were not randomized to drug or placebo if they withdrew consent, were unable to complete baseline procedures or no longer met inclusion criteria.
Period: Overall Study
Arm/Group | Simvastatin | Placebo
Started | 44 | 44
Completed | 42 | 41
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — withdrew from study due to busy schedule | 1 | 1
Not completed — Mental health issues | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Simvastatin | Placebo | Total
Number analyzed (Participants) | 44 | 44 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 38 | 79
  >=65 years | 3 | 6 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.95 (6.2) | 54.4 (7.8) | 55.21 (6.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 32 | 63
  Male | 13 | 12 | 25
Region of Enrollment [Number; unit: participants]
  United States | 44 | 44 | 88

OUTCOME MEASURES:

1. Primary Outcome: Changes in Cerebrospinal Fluid (CSF) Beta-amyloid-42 Levels Compared to Baseline as Measured by xMAP
Description: Change in CSF beta-amyloid-42 was defined as the ratio of 18-month levels to baseline levels.
  Beta-amyloid-42 is a substance found in the plaques in the brain of people with Alzheimer's disease and can be detected in CSF. There is no defined normal range yet for middle-aged adults.
Time Frame: Baseline and 18 months
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 39 | 40
ratio | 1.01 [0.96 to 1.07] | 0.98 [0.95 to 1.02]

2. Secondary Outcome: Changes in CSF Beta-amyloid-40 Levels as Measured by xMAP (Multi-Analyte Profiling) )
Description: Change in CSF beta-amyloid-40 was defined as the ratio of 18-month levels to baseline levels.
  Beta amyloid-40 is a substance found in the brain vessels of individuals with Alzheimer's disease and has more potent cerebrovascular effects on individuals with Alzheimer's disease than any other form of beta amyloid.
Time Frame: Baseline and 18 months
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 39 | 40
ratio | 1.03 [0.99 to 1.07] | 0.98 [0.94 to 1.01]

3. Secondary Outcome: Changes in CSF Soluble Alpha Precursor Proteins (sAPP-alpha) and Soluble Beta Precursor Proteins (sAPP-beta) as Measured by Duplex
Description: Changes in CSF sAPP-alpha and sAPP-beta were defined as the ratio of 18-month levels to baseline levels.
  sAPP-alpha and sAPP-beta are components of beta-amyloid that provide information on beta-amyloid breakdown.
Time Frame: Baseline and 18 months
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 39 | 40
ratio
  sAPP-alpha | 0.96 [0.92 to 1.00] | 1.03 [0.97 to 1.09]
  sAPP-beta | 0.98 [0.93 to 1.02] | 1.00 [0.97 to 1.04]

4. Secondary Outcome: Changes in CSF Total Tau (T-tau) and Phosphorylated Tau (P-tau) as Measured by xMAP
Description: Changes in CSF t-tau and p-tau were defined as the ratio of 18-month levels to baseline levels.
  T-tau and p-tau are substances found in the brain that can provide information on nerve cell health in the brain and tangle formation in nerve cells.
Time Frame: Baseline and 18 months
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 39 | 40
ratio
  Total tau | 1.01 [0.97 to 1.05] | 1.01 [0.98 to 1.05]
  Phosphorylated tau | 1.16 [0.90 to 1.42] | 1.15 [1.00 to 1.29]

ADVERSE EVENTS:
Arm/Group | Simvastatin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 0/44 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes